CLINICAL TRIAL: NCT05582837
Title: Treatment of Meniere's Disease With Nortriptyline-Topiramate Stepwise Regimen: A Randomized Double-Blinded Clinical Trial
Brief Title: Treatment of Meniere's Disease With Migraine Medications
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Hamid Djalilian, Professor, Neurotology and skull base surgery, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20216445
Record Dates: First submitted 2021-10-07; First posted 2022-10-17 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Ménière
Keywords: Meniere's Disease, medication, randomized, trial, migraine
MeSH Terms: conditions — Meniere Disease; Migraine Disorders | interventions — Nortriptyline; Topiramate

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to a study group by chance (like a coin flip) rather than by a medical decision made by the researchers. There are two arms in the study (treatment group which consists of nortriptyline + topiramate, control group which consist of hydrochlorothiazide plus triamterene with placebo), and participants enrolling in the trial will be randomly assigned in a 1:1 fashion to one of the arms. The participant will remain in the same arm for the duration of the study (8 weeks). There may be multiple participants in each arm who are undergoing the study at the same time (parallel model).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: No masking: care provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- nortriptyline + topiramate (Experimental): Nortriptyline (starting dose 7.5 mg) plus Topiramate (starting dose 10 mg) with appropriate dosage increase as necessary
  Interventions: Drug: nortriptyline + topiramate
- hydrochlorothiazide + triamterene + placebo (Active Comparator): hydrochlorothiazide (starting dose 25 mg) plus triamterene (starting dose 37.5 mg) with placebo being added in case of a dosage increase
  Interventions: Drug: nortriptyline + topiramate

INTERVENTIONS:
Drug: nortriptyline + topiramate — nortriptyline (7.5mg) + topiramate (10mg) taken 1x per day and escalate weekly as needed for 8 weeks
  Other Names: Pamelor, Topamax

SUMMARY:
Meniere's disease (MD) is a chronic disease with a variety of fluctuating signs and symptoms, which include vertigo, hearing loss, tinnitus (ringing noise in the ear), aural pressure (feeling of ear fullness), and disequilibrium (lack of stability). Vertigo represents one of the most common and distressing problems in MD patients, and it causes various somatic and psychological disorders that interfere with the patient's quality of life. Despite the large economic and emotional impact of symptoms in MD patients, there is no FDA-approved medication to treat this debilitating condition. As such, our objective in this study is to evaluate the therapeutic potential of novel medications in treating MD that have previously shown astonishing promise in our clinical practice.

DETAILED DESCRIPTION:
This study is 8 weeks in duration. There are two arms in the experiment: the first is nortriptyline (7.5 mg) plus topiramate (10 mg), the second is hydrochlorothiazide (25 mg) plus triamterene (37.5 mg) with placebo being added in case of a dosage increase. This is a double-blinded trial. Participants will be randomized to one arm for the duration of the trial using simple randomization with a computer-generated number. Both groups may receive dosage increases weekly if symptoms do not improve. Symptomatic survey scores from each arm will be obtained before and after treatment and weekly. An unblinded clinical researcher will also become involved with patients' treatments as they start to report changes in symptoms in order to monitor their safety and provide advice on change in dosage if patients have questions.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with active or frequent Meniere's Disease.
2. Male or female between the ages of 25 to 85 years.
3. Subject must be compliant with the medication and attend study visits.
4. Must be able to read and write in the English language to provide consenting.

Exclusion Criteria:

1. Pregnancy will result in automatic exclusion from the study. A urine pregnancy test to rule out pregnancy for all women who are of childbearing potential.
2. Subjects with history of surgery for Meniere's Disease.
3. Subject with history of an adverse reaction to medication being prescribed.
4. Subject suffers from a medical condition or has history that may be concerning to the investigator's clinical opinion.
5. Subjects with psychosis.
6. Subjects with neurological neoplasm.
7. All contraindications for the medications which prevent subjects from randomization will be considered as exclusion criteria.

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Subjective improvement of Meniere's Disease | 8 weeks
  The primary outcome variable is derived from the validated Meniere's Disease Outcome Questionnaire (MDOQ) with 18 multiple-choice questions to compare quality of life before and after treatment. The question multiple choices are rated on a scale from 0 to 4 where the higher score indicates the higher quality of life. For each patient, the sum of his/her answers is divided (and x100) by the maximum possible scores for the pre-treatment questions and the post-treatment questions, separately. The outcome measure is the absolute change from pre- to post-treatment scores. Two-sample t test will be used to compare the outcome variable between the two treatment groups.

SECONDARY OUTCOMES:
Visual analog scale (VAS) | 8 weeks
  Subjective improvement in tinnitus loudness severity based on a visual analog scale (VAS). The VAS is scored from 0 to 10, with a higher score representing an increased severity of tinnitus.
Perceived Stress Scale (PSS) | 8 weeks
  Subjective improvement in stress based on perceived stress scale (PSS). The PSS is scored from 0 to 40, with higher scores indicating higher perceived stress.
Sleep Quality Index (SQI) | 8 weeks
  Subjective improvement in sleep quality based on sleep quality index (SQI). The SQI is scored from 0 to 21, with higher scores indicating worse quality of sleep.
Dizziness handicap index (DHI) | 8 weeks
  Subjective improvement in dizziness handicap index (DHI). There is a maximum score of 100 (28 points for physical, 36 points for emotional and 36 points for functional) and a minimum score of 0. The higher the score, the greater the perceived handicap due to dizziness.
Tinnitus Functional Index (TFI) | 8 weeks
  Subjective improvement from baseline in tinnitus symptoms as measured by Tinnitus Functional Index (TFI). The TFI is scored from 0% to 100%, with higher scores indicating a more negative impact of tinnitus.
Meniere's Disease Outcomes Questionnaire (MDOQ) | 8 weeks
  Subjective improvement in Meniere's Disease Outcomes Questionnaire (MDOQ). To measure the quality of life in patients with Ménière's disease and to assess quality-of-life outcomes.
Patient Health Questionnaire (PHQ) | 8 weeks
  Subjective improvement in depression symptoms based on patient health questionnaire (PHQ). The PHQ is scored from 0 to 27, with a higher score indicating increased depression severity.

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Djalilian, MD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine Medical Center ENT Clinic (Pavilion 2), Orange, California, United States